CLINICAL TRIAL: NCT03165695
Title: Ramelteon vs Placebo for Prevention of Delirium and Improvement of Sleep in Hospitalized Older Adults
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Never funded
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Elizabeth B. Klerman, Associate Professor of Medicine, Harvard Medical School, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2017P000656
Record Dates: First submitted 2017-05-22; First posted 2017-05-24 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Delirium in Old Age
Keywords: Delirium; Insomnia; Ramelteon
MeSH Terms: conditions — Delirium; Sleep Initiation and Maintenance Disorders | interventions — ramelteon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ramelteon Arm (Experimental): Ramelteon tablet 8 mg orally at 21:00 for 7 days or until discharge whichever comes first.
  Interventions: Drug: Ramelteon
- Placebo Arm (Placebo Comparator): Sugar pill manufactured to mimic Ramelteon 8 mg tablet orally at 21:00 for 7 days or until discharge whichever comes first.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ramelteon — Ramelteon 8 mg tablet orally at 21:00 for 7 days or until discharge whichever comes first
  Other Names: Rozerem
  Arms: Ramelteon Arm
Drug: Placebo — Placebo, 1 tablet orally at 21:00 or until discharge whichever comes first
  Arms: Placebo Arm

SUMMARY:
This study evaluates whether Ramelteon can prevent delirium, decrease the severity of incident delirium and improve sleep wake cycle in hospitalized elderly surgical patients. Half of the patients will be assigned to Ramelteon, while other half will be assigned to placebo.

DETAILED DESCRIPTION:
Delirium is a common clinical syndrome characterized by acute cognitive dysfunction with core features of inattention, disorganized thinking, perceptual disturbances and sleep-wake cycle disruption. It is typically multifactorial and can be triggered by acute infection, metabolic derangements, surgery, and certain medications. Older adults have a much higher incidence of delirium. Delirium increases in-hospital mortality, length of stay, rate of institutionalization and may cause or exacerbate cognitive impairment. The present pilot study investigates sleep loss as potentially important contributing factors in delirium and an opportunity for intervention. Sleep disruption is prevalent among hospitalized patients. Sufficient sleep is important for recovery from illness, management of pain, wound healing, and a variety of other biologic functions integral to recovery in addition to its putative role in delirium prevention. Melatonin plays an important role in circadian rhythms and sleep-wake cycle regulation. Melatonin secretion is altered in hospitalized older patients in comparison with community-living older individuals. Melatonin and the melatonin-receptor agonist Ramelteon have been studied and have shown promise in delirium prevention, in addition to promoting sleep. We propose to test the use of Ramelteon to decrease delirium and improve sleep/wake cycles in the elderly surgical patients.

ELIGIBILITY:
Inclusion Criteria:

* 65 years of age or older.
* Admitted to BWH vascular surgical service.
* Able to provide informed consent or a surrogate is available to provide informed consent.
* Absence of delirium at time of consent.

Exclusion Criteria:

* Expected stay or life expectancy less than 48 hours
* Unable to take medications orally
* Advanced liver disease (Child-Pugh class B or worse)
* Active treatment with Fluvoxamine
* Active treatment with antipsychotic medications, benzodiazepines or other hypnotic agents (i.e. Trazodone, Mirtazapine, Zolpidem, Zaleplon)
* Known or suspected diagnosis of Lewy body dementia
* Any dermatological condition that may be aggravated by using a wrist sensor.
* Known pre-existing sleep disorder other than insomnia.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of delirium | 7 days or less depending on the length of hospital stay
  Incidence of delirium measured by DRS-98R

SECONDARY OUTCOMES:
Severity of delirium | 7 days or less depending on the length of hospital stay
  Decreased mean DRS-98R score
Sleep improvement | 7 days or less depending on the length of hospital stay
  Improvement in sleep metrics: increased duration of sleep as measured by Actigraphy

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth B Klerman, M.D.,PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No